CLINICAL TRIAL: NCT06965855
Title: Revolution or Routine? Assessing the Postoperative Impact of Piezoelectric Surgery on Edema, Trismus, and Other Complications in Third Molar Extractions
Brief Title: Effect of Piezoelectric Surgery onPostoperative Complications in Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mert Zeytinoğlu, Assoc. Prof. Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EGE-DHF-MZ-003
Record Dates: First submitted 2025-04-25; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Oral Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 patients in the piezoelectric surgery group (Experimental)
  Interventions: Procedure: piezoelectric surgery
- 30 patients in the conventional surgery group (Experimental)
  Interventions: Procedure: conventional surgery

INTERVENTIONS:
Procedure: conventional surgery — This retrospective clinical study included 30 patients who underwent extraction of impacted lower third molars with conventional surgery
  Arms: 30 patients in the conventional surgery group
Procedure: piezoelectric surgery — Description: This retrospective clinical study included 30 patients who underwent extraction of impacted lower third molars with piezoelectric surgery
  Arms: 30 patients in the piezoelectric surgery group

SUMMARY:
The purpose of this study is to compare the effects of piezoelectric surgery on postoperative edema, trismus and other postoperative complications (Wound Healing, Bleeding, Infection, Alveolitis, Paresthesia) with conventional bur method applied in surgical extraction of impacted mandibular third molars.

The main question it aims to answer is:

Is piezoelectric surgery effective on reducing the edema, trismus and other postoperative complications (Wound Healing, Bleeding, Infection, Alveolitis, Paresthesia) in impacted third molar surgery? Postoperative edema measurements are determined at 24 hours, 48 hours, and 7 days using the flexible ruler method. Trismus is determined by measuring the interincisal distance. Statistical analyses are performed to compare the two surgical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mesioangular, distoangular, vertical or horizontal, fully impacted and fully bone retained impacted lower wisdom teeth
* Patients without any systemic disease
* Patients who have been informed about the duration, purpose and requirements of the study and who have signed the informed consent form voluntarily.

Exclusion Criteria:

* Patients with any systemic contraindication, infection in the area of the tooth to be extracted, anamnesis of sensitivity to paracetamol derivatives or aspirin, pregnant or breastfeeding patients, and patients using antibiotics or anti-inflammatory drugs in the last 3 weeks
* In addition, smokers or alcohol addicts were not included in the study.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2013-01-01 (Actual)

PRIMARY OUTCOMES:
Edema amounts with Routine and Piezoelectric Surgery | The edema measurements are made on the patient preoperatively and on the 2nd and 7th postoperative days.
  Edema measurements are made on the distances between the corner of the eye and the angulus mandible, between the tragus and the corner of the mouth, and between the tragus and the soft tissue pogonium. These points were marked with a dermatological pen and measured with the flexible ruler method.
Trismus amounts with Routine and Piezoelectric Surgery | The trismus measurements are made on the patient preoperatively and on the 2nd and 7th postoperative days.
  In order to determine the trismus, the values of the mouth openings of the patients are obtained by measuring the distance between the mesial corners of the first permanent incisors in the upper and lower jaws with the help of a caliper (Mitutoyo Company, Japan) with a sensitivity of 0.05.

SECONDARY OUTCOMES:
Wound healing, bleeding, infection, alveolitis, paresthesia, and temporomandibular joint pain with Routine and Piezoelectric Surgery | within 7 days after surgery
  These complications are recorded by clinical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Mert Zeytinoğlu, Principal Investigator — Ege University

IPD SHARING:
Plan to Share IPD: No